CLINICAL TRIAL: NCT02200757
Title: A Multicenter, Randomized, Open-Label Phase 2b Study to Investigate the Efficacy and Safety of Aldoxorubicin Compared to Topotecan in Subjects With Metastatic Small Cell Lung Cancer Who Either Relapsed or Were Refractory to Prior Chemotherapy
Brief Title: Efficacy and Safety of Aldoxorubicin Compared to Topotecan in Subjects With Metastatic Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALDOXORUBICIN-P2-SCLC-01
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2016-01

CONDITIONS: Metastatic Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — DOXO-EMCH; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aldoxorubicin (Experimental)
  Interventions: Drug: Aldoxorubicin
- Topotecan (Active Comparator)
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Aldoxorubicin — 230 mg/m2 (170 mg/m2 doxorubicin equivalent) intravenously on Day 1 of each 21-day cycle. Number of cycles: until tumor progression or unacceptable toxicity occurs.
  Other Names: INNO-206
  Arms: Aldoxorubicin
Drug: Topotecan — 1.5 mg/m2/day intravenously for 5 consecutive days on Day 1 of each 21-day cycle OR 4 mg/m2 intravenously on Days 1, 8 and 15 of each 28-day cycle. Number of cycles: until tumor progression or unacceptable toxicity occurs
  Other Names: Hycamtin
  Arms: Topotecan

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of aldoxorubicin compared to topotecan in subjects with metastatic small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years male or female.
2. Histological confirmation of SCLC.
3. Relapsed or refractory to no more than 1 course of a systemic therapy regimen and is incurable by either surgery or radiation.
4. Capable of providing informed consent and complying with trial procedures.
5. ECOG PS 0-2.
6. Life expectancy >8 weeks.
7. Measurable tumor lesions according to RECIST 1.1 criteria.[22]
8. Women must not be able to become pregnant (e.g. post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. (Adequate contraception includes: oral contraception, implanted contraception, intrauterine device implanted for at least 3 months, or barrier method in conjunction with spermicide.)
9. Males and their female partner(s) of child-bearing potential must use 2 forms of effective contraception (see Inclusion 8 plus condom or vasectomy for males) from the last menstrual period of the female partner during the study treatment and for 6 months after the final dose of study treatment.
10. Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
11. Accessibility to the site that ensures the subject will be able to keep all study-related appointments.

Exclusion Criteria:

1. Prior exposure to >375 mg/m2 of doxorubicin or liposomal doxorubicin.
2. Prior treatment with topotecan.
3. Palliative surgery and/or radiation treatment < 21 days prior to date of randomization.
4. Exposure to any investigational agent within 30 days of date of randomization.
5. Exposure to any systemic chemotherapy within 21 days of date of randomization.
6. Active (symptomatic) central nervous system (CNS) metastasis.
7. History of other malignancies except cured basal cell carcinoma, cutaneous squamous cell carcinoma, melanoma in situ, superficial bladder cancer or carcinoma in situ of the cervix unless documented free of cancer for ≥3 years.
8. Laboratory values: Screening serum creatinine >1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) >3×ULN or >5×ULN if liver metastases are present, total bilirubin >2×ULN, absolute neutrophil count (ANC) <1,500/mm3, platelet concentration <100,000/mm3, hemoglobin <9 g/dL, albumin <2 gm/dL.
9. Anion gap > 16 meq/L or arterial blood pH < 7.30.
10. Clinically evident congestive heart failure (CHF) > class II of the New York Heart Association (NYHA) guidelines (Appendix D).
11. Current, serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V (Appendix F).
12. Baseline QTc >470 msec measured by Fridericia's formula (QTcF) and/or previous history of QT prolongation while taking other medications. Concomitant use of medications associated with a high incidence of QT prolongation is not allowed.
13. History or signs of active coronary artery disease with angina pectoris within the last 6 months.
14. Serious myocardial dysfunction defined by ECHO as absolute left ventricular ejection fraction (LVEF) below the institution's lower limit of predicted normal.
15. Known history of HIV infection.
16. Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals.
17. Treatment with p-glycoprotein inhibitors such as cyclosporine A, elacridar, ketoconazole, ritonavir, saquinavir.
18. Major surgery within 30 days prior to date of randomization.
19. Substance abuse or any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
20. Any condition that is unstable and could jeopardize the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - City of Hope Medical Group, Pasadena, California
  - Cancer Specialists of North Florida-Fleming Island, Fleming Island, Florida
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Oncology Hermatology Care, Inc., Cincinnati, Ohio
  - Northwest CCOP Kaiser Permanente, Portland, Oregon
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Hungary (6):
  - Koranyi National Institute of TBC and Pulmonologyhhy, Budapest
  - Koranyi National Institute of TBC and Pulmonology, Budapest
  - University of Debrecen, Medical and Health Science Center, Department of Pulmonology, Debrecen
  - Szabolcs-Szatmar-Bereg County Hospitals and University Teaching Hospital, Department of Pulmonology, Nyíregyháza
  - Medical Center of the University of Pecs, 1st Department of Internal Medicine, Pécs
  - Hetenyi Geza Hospital, Szolnok
- Spain (12):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Quiron-Dexeus (IOR), Barcelona
  - University Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Lucus Augusti, Lugo
  - General University Hospital Gregorio Maranon, Madrid
  - Hospital Puerta de Hierro, Madrid
  - University Hospital Foundation Jimenez Diaz, Madrid
  - University Hospital La Paz, Madrid
  - Hospital Regional Universitario, Málaga
  - University Hospital Virgen de Valme, Seville
  - CHU Xeral, Vigo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 135 subjects were enrolled in the intent to treat population, whereas 130 subjects were in the safety population.
  5 subjects were discontinued prior to treatment start.
Groups:
- Aldoxorubicin: Aldoxorubicin: 230 mg/m^2 (170 mg/m^2 doxorubicin equivalent) intravenously on Day 1 of each 21-day cycle. Number of cycles: until tumor progression or unacceptable toxicity occurs.
- Topotecan: Topotecan: 1.5 mg/m^2/day intravenously for 5 consecutive days on Day 1 of each 21-day cycle OR 4 mg/m^2 intravenously on Days 1, 8 and 15 of each 28-day cycle. Number of cycles: until tumor progression or unacceptable toxicity occurs
Period: Overall Study
Arm/Group | Aldoxorubicin | Topotecan
Started | 67 | 63
Completed | 67 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2 subjects were randomized, but not treated in the Aldoxorubicin Arm. 3 subjects were randomized, but not treated in the Topotecan Arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aldoxorubicin | Topotecan | Total
Number analyzed (Participants) | 69 | 66 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (6.73) | 63.5 (7.72) | 64.42 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 26 | 60
  Male | 35 | 40 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 61 | 56 | 117
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 64 | 62 | 126
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Subjects with Metastatic Small Cell Lung Cancer [Count of Participants; unit: Participants] | 69 | 66 | 135

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to first documentation of objective tumor progression or to death due to any cause in the absence of previous documentation of objective tumor progression.
  Progressive Disease is defined as: ≥20% increase in the sum of the longest diameter of target lesions from the smallest sum of the longest diameter recorded since the treatment started; the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of ≥1 new lesion is also considered progression.
Time Frame: 24 months
Population: PFS is measured from randomization, not from treatment start date. 2 subjects were randomized, but not treated in the Aldoxorubicin Arm. 3 subjects were randomized, but not treated in the Topotecan Arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Aldoxorubicin | Topotecan
Number analyzed (Participants) | 69 | 66
Months | 1.5 [1.4 to 2.7] | 2.7 [1.5 to 3.0]

2. Secondary Outcome: Number of Participants With Treatment-related Toxicities (Adverse Events)
Time Frame: Treatment was planned to continue until tumor progression is observed, subject asks to withdraw, or unacceptable toxicity occurs, up to 451 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Aldoxorubicin | Topotecan
Number analyzed (Participants) | 67 | 63
Participants | 51 | 52

ADVERSE EVENTS:
Time Frame: All AEs and SAEs that occurred after any administration of the study medication were to be followed until the event resolved, until the subject began alternative treatment, or until 30 days after the last dose of study medication, up to 451 days.
Description: 2 subjects were randomized, but not treated in the Aldoxorubicin Arm. 3 subjects were randomized, but not treated in the Topotecan Arm.
  135 subjects were enrolled in the intent to treat population, whereas 130 subjects were in the safety population.
  5 subjects were discontinued prior to treatment start.
  Mortality was assessed in all enrolled subjects. AEs/SAEs were assessed in the safety population, all patients who received at least one dose of any study drug.
Arm/Group | Aldoxorubicin | Topotecan
All-Cause Mortality (participants affected / at risk) | 57/69 | 50/66
Serious Adverse Events (participants affected / at risk) | 17/67 | 18/63
Other Adverse Events (participants affected / at risk) | 61/67 | 61/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldoxorubicin (N=67) | Topotecan (N=63)
Pneumonia (Infections and infestations) | 3 | 2
Respiratory tract infection (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypomobility (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aldoxorubicin (N=67) | Topotecan (N=63)
Anaemia (Blood and lymphatic system disorders) | 16 | 25
Neutropenia (Blood and lymphatic system disorders) | 12 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 30
Leukopenia (Blood and lymphatic system disorders) | 2 | 4
Lymphopenia (Blood and lymphatic system disorders) | 4 | 2
Fatigue (General disorders) | 14 | 13
Asthenia (General disorders) | 10 | 15
Chest pain (General disorders) | 2 | 4
Gait disturbance (General disorders) | 2 | 4
Oedema peripheral (General disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 12 | 11
Constipation (Gastrointestinal disorders) | 9 | 9
Stomatitis (Gastrointestinal disorders) | 13 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 9
Vomiting (Gastrointestinal disorders) | 7 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 12 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 4 | 3
Pneumonia (Infections and infestations) | 4 | 2
Respiratory tract infection (Infections and infestations) | 4 | 2
Bronchitis (Infections and infestations) | 4 | 1
Headache (Nervous system disorders) | 7 | 2
Dizziness (Nervous system disorders) | 2 | 6
Dysgeusia (Nervous system disorders) | 2 | 4
Platelet count decreased (Investigations) | 4 | 10
Neutrophil count decreased (Investigations) | 7 | 4
White blood cell count decreased (Investigations) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT02200757/Prot_SAP_000.pdf